CLINICAL TRIAL: NCT00249639
Title: Contingency Management for Attendance
Brief Title: Contingency Management for Attendance - 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: UConn Health (Other)
Responsible Party: Nancy Petry, Ph.D., UConn Health Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-16855-2; R01-16855-2
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-05

CONDITIONS: Substance Abuse
Keywords: Contingency Management; Substance Abuse Treatment
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Contingency management — Rewards valued $1-$100

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a low-cost contingency management procedure as compared to standard treatment. Using a cross-over design, CM is implemented at different community-based clinics and compared with non-CM in the same facilities. Research staff collects information regarding patients' demographic characteristics, attendance, and outcomes at the clinics. During Phase A (non-CM), standard clinical practice is in place. During Phase B (CM), all patients have the chance to win prizes by coming to treatment. Each participating clinic is randomly assigned to receive either the A or B phase first; each phase is in effect for 16 weeks.

ELIGIBILITY:
Subjects will be patients in treatment at one of the participating clinics during the study period. There are no other inclusion or exclusion criteria because we wish to make enrollment open to increase generalizability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2004-01; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Drug use | baseline and each follow-up
Retention | baseline and each follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Petry, Ph.D., Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States